CLINICAL TRIAL: NCT06039618
Title: Capabilities of Perinatal Healthcare Institutions in Primary and Tertiary Care of Low Birth Weight Infants in the Federation of Bosnia and Herzegovina: A Cross-sectional Multicentric Study.
Brief Title: Capabilities of Perinatal Healthcare Institutions in the Federation of Bosnia and Herzegovina
Status: Completed | Type: Observational
Sponsor: Evangelisches Krankenhaus Bethesda zu Duisburg (Other)
Responsible Party: Principal Investigator, Antoine Naem, Research Assistant, Evangelisches Krankenhaus Bethesda zu Duisburg
Other Study IDs: 02-09/2-77/20
Record Dates: First submitted 2023-09-06; First posted 2023-09-15 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Prenatal Care

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Referred to a Centre of Higher Level: Those are the newborns that were referred at the time of delivery or within one week after birth to centers of higher organizational level.
  Interventions: Other: Referral to Centre of Higher Organizational Level
- Treated at the Centre of Admission: Those are the newborns that were not referred to other centers and were treated in the health facility were the birth took place, and hospitalized in the same center until discharge.

INTERVENTIONS:
Other: Referral to Centre of Higher Organizational Level — Referral to Centre of Higher Organizational Level. This means referral from a primary neonatal care center to a secondary one, or from the secondary to the tertiary center.
  Groups: Referred to a Centre of Higher Level

SUMMARY:
The aim of this study is to assess the level of the perinatal healthcare institution (PHI) where the newborns were delivered. We included newborns of both genders that were born in the maternity wards in 10 cantons of the Federation of Bosnia and Herzegovina (FBiH). From the PHI of the first and second level, 159 newborns were referred to the third level. Out of a total of 159 LBWI referred from other PHI, only 19.5% LBWI were transported in less than 4 hours. In second level PHI, most LBWI died in the first 12 hours after birth.

ELIGIBILITY:
Inclusion Criteria:

* Newborns of both genders that were born in the maternity wards in 10 cantons of the FBiH
* A gestational age between 22 and 42 weeks, and a birth weight less than 2500g.

Exclusion Criteria:

* Infants younger than 22 weeks or older than 42 weeks.
* Infants whose mothers refused to give consent for participation in the study.

Ages: 22 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Newborns that were born in the maternity wards of the Federation of Bosnia and Herzegovina
Sampling Method: Non-Probability Sample
Enrollment: 22897 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Referral to a centre of higher organizational level. | Before birth and up to 4 hours or more after delivery.
  Referring the neonate with low birth weight to a more specialized centre.

CONTACTS AND LOCATIONS:
Overall Officials: Anis Cerovac, M.D., Principal Investigator — General Hospital Tešanj
Locations (1):
- General Hospital Tešanj, Tešanj, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: No